CLINICAL TRIAL: NCT06399016
Title: The Effect of Reading a Book With Augmented Reality Application on the Level of Fear and Anxiety in Children in the 7-12 Age Group in the Preoperative Period
Brief Title: Augmented Reality Applied Book Reading in the Preoperative Period
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Duygu Karaarslan, Assistant professor, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Augmented Reality Application
Record Dates: First submitted 2024-04-28; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Preoperative Anxiety
Keywords: Child; fear; anxiety; operating theater tour; augmented reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: During the preoperative period, children who meet the inclusion criteria of the study will be determined from the list of children who will undergo surgery. Before the research, children who will undergo surgery and their parents will be informed on the morning of the surgery, approximately 1 hour before the surgery, and their written and verbal consent will be obtained. On the morning of the surgery day, the "Child and Family Introductory Data Form" will be filled out by children in the 7-12 age group and their parents who meet the inclusion criteria and agree to participate in the research. The child himself/herself will be asked to score the level of surgery-related anxiety using the "CAS" score, and the child, the parent, and the researcher will be asked to score the child's fear level regarding the surgery using the "CFS" score.
  The application material to be used in the research is the story book titled 'One Child, One Miracle', which includes an augmented reality application.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the process of assignment of children into groups, randomization is achieved in the computer by stratifying them in terms of sex and age variables (https://www.randomizer.org/).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Augmented Reality Applied Book Reading Group (Experimental): Children included in this group will be asked to read books supported by augmented reality technology. Approximately 1 hour before the surgery, a survey will be administered to the child and the accompanying parent using the "Child and Family Introductory Data Form", which includes sociodemographic characteristics. The child himself/herself will be asked to score the level of surgery-related anxiety using the "CAS" score, and the child, the parent, and the researcher will be asked to score the child's fear level regarding the surgery using the "CFS" score. Data collection will take approximately 10 minutes in total. Immediately afterwards, the researcher will ask the child to read the book 'One Child, One Miracle', which is a technology-supported augmented reality application, with the help of an application previously downloaded free of charge from Google Play or IOS to a mobile phone or tablet.
  Interventions: Device: augmented reality book
- Group 2: Control Group (Experimental): In the preoperative period, the researcher will conduct a survey on the morning of the surgery day, approximately 1 hour before the surgery, using the "Child and Family Introductory Data Form", which includes the sociodemographic characteristics of the child and the accompanying parent. The child himself/herself will be asked to score the level of surgery-related anxiety using the "CAS" score, and the child, the parent, and the researcher will be asked to score the child's fear level regarding the surgery using the "CFS" score. Data collection will take approximately 10 minutes in total. Immediately afterwards, the child will be asked by the researcher to read the story book "One Child, One Miracle". This group will be asked to just read the book without turning on the book's augmented reality feature. Afterwards, using the same scales, children will score the "CAS" scales, and the child, parent and researcher will score the "CFS" scales.
  Interventions: Device: book

INTERVENTIONS:
Device: augmented reality book — The story will be presented to the children in this application group in three dimensions. The augmented reality application will be supported by the researcher as it must be used under the supervision of an adult. When the tablet or phone is held to the pages of the book, the animations of these pages are displayed on the screen with sound. While the animation opens automatically when we hold the phone or tablet, the story can be listened to aloud at the same time.
  Other Names: Augmented reality applied book titled 'One Child, One Miracle'
  Arms: Group 1: Augmented Reality Applied Book Reading Group
Device: book — This group will be asked to just read the book without turning on the augmented reality feature of the book.
  Other Names: 'One Child, One Miracle'
  Arms: Group 2: Control Group

SUMMARY:
Non-pharmacological methods such as multimedia applications and visual and auditory technological tools are used to create a more enjoyable experience by reducing children's fear and anxiety and distracting them in the preoperative period. With the latest developments in technology, live, immersive, augmented and virtual reality systems are seen to be included and used in preoperative preparation training, especially for pediatric patients. One of the applications of these innovative technologies that has attracted attention recently is augmented reality technology. The original value of this study is to reduce the fear and anxiety levels experienced by children reading books in the preoperative period with the application of augmented reality, which is a developing, promising and easily accessible technology. The method of this study consists of two groups: an augmented reality applied book reading group and a control group. In the preoperative period for both groups, a survey will be administered to the child and the accompanying parent using the "Child and Family Introductory Data Form", which includes sociodemographic characteristics, approximately 1 hour before the surgery. In addition, the child himself will be asked to score the "Child Anxiety Scale-State" scale to determine the level of anxiety about the surgery, and the child himself, the parent and the researcher will be asked to score the "Child Fear Scale" to determine the child's level of fear about the surgery. The book reading group with augmented reality application will be asked to read the voiced and animated book titled 'One Child, One Miracle', accompanied by an application downloaded free of charge from Google Play or IOS to their mobile phone or tablet. The storybook will be presented to the children in this application group in three dimensions with the help of a mobile phone or tablet. Children in the control group will read the same book without using the augmented reality application. After reading the book for both groups, the children will be asked to rate their fear and anxiety levels again using the same scales. This research is a randomized controlled and experimental study. The adequacy of the sample size in the study "G. It was calculated using the "Power-3.1.9.2" program. In the power analysis conducted for the sample and power calculation of the experimental study with the application and control groups, it was decided to study with 30 children for each group.

DETAILED DESCRIPTION:
During hospitalization and exposure to medical procedures and surgical procedures, children perceive themselves as different from other children and experience feelings of inadequacy and feel hindered. Especially for school-age children aged 7-12, hospitalization means a process full of worries that cause anxiety and fear. In a study investigating the feelings of hospitalized children aged 7-12 about "hospital" and "disease", it was observed that children defined the hospital as a place where pain and painful procedures are performed most often, causing both themselves and their parents to be upset, and where they experience fear and anxiety. Because the hospital environment, staff, materials used and procedures to be performed are reflected as a state of uncertainty for every group of children hospitalized. This uncertainty they experience may affect the child's adaptation to the hospital and treatment, his communication with healthcare personnel, and his future hospital experience. Having an additional surgical intervention on the child in addition to hospitalization causes more stress and affects the child more both psychologically and physiologically. In a study, the psychosocial symptoms of 360 hospitalized children aged 6-12 were examined in terms of some variables. It has been determined that more than half of the children develop "anxiety" due to hospitalization, along with "regression", "communication difficulty", "hopelessness" and "anger" behaviors. In another study examining postoperative behavioral changes in Chinese children who underwent hypospadias surgery, it was determined that three-fifths of the children showed behavioral changes that lasted for several weeks after surgery.

The success of surgery in children is not only related to the importance of the techniques and skills applied, but also to the preparation of the child and the parent and meeting the care needs in the preoperative period. Preparing the child patient appropriately in the preoperative period prevents him from experiencing both behavioral and physiological symptoms of fear and anxiety. Studies have shown that more than 60% of children who undergo surgery experience anxiety before surgery and anesthesia. However, in children who were psychologically affected in the preoperative period, maladaptive behavioral changes such as anxiety, eating and sleeping disorders, nightmares, enuresis and tantrums occurred in the postoperative period. Some intervention practices have been developed to reduce preoperative fear and anxiety in children and to prevent anxiety-related behavioral changes. These practices include various behavioral preparation programs used to distract from nonpharmacological practices. Such approaches help children to divert their attention from fearful and painful procedures by keeping them active. In methods of diverting attention; Methods such as daydreaming, listening to music, hypnosis, relaxation techniques, breathing control, biofeedback exercises, watching videos, reading books, telling stories and games are used. In a study, it was observed that children aged 4-10 years of age reduced their stress, their parents' anxiety, and postoperative delirium by providing distraction via tablets and phones in the preoperative period, and increased cooperation with medical personnel during anesthesia induction. The preparations to be made according to the child's age, period characteristics and understanding capacity should be explained to the child so that he/she does not feel afraid. Because preoperative anxiety is associated with an increased incidence of delirium, pain, and postoperative maladaptive behavior in the child. It can also manifest itself in various ways such as agitation, crying, shaking, struggle and escape behaviors. Therefore, the main goal in preparing for the surgery process is to maintain the child-parent relationship, reduce fears and anxiety arising from the unknown, and psychologically support the child and parents. Preoperative interventions have been increasingly used in hospital settings over the past few years. It has been observed that fear and anxiety arising from the preoperative period in children, video glasses, video displaying smartphones and tablets reduce postoperative delirium.

Hypothesis of the Research:

Hypothesis 1. H1: Reading books with augmented reality application in the preoperative period reduces the level of fear in children aged 7-12.

Hypothesis 2. H1: Reading books with augmented reality application in the preoperative period reduces the anxiety level in children aged 7-12.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7-12
* Children who will undergo surgery for the first time will be included
* No communication problems (vision, hearing, mental),
* Both his/her parents volunteer to participate in the research, and their parents give written and verbal consent,

Exclusion Criteria:

* Children have genetic or congenital disease,
* Children have a chronic disease
* Children have previous surgery

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Information Form | in the preoperative period.
  A total of 23 questions are the researcher prepared the form in line with the literature.
  The form is include two parts. One of theparts are include items questioning the child's diagnosis, length of hospital stay, sex, and whether he or she had been hospitalized or had surgery previously. The forms will filled by the researcherusing the face-to-face interview method.

SECONDARY OUTCOMES:
Determining the preoperative anxiety scores of children | in the preoperative period.
  This scale is a one-item self-report measure for measuring fear in level of children aged 5-12 years. Psychometric properties of Child fear scale in Turkish population were conducted by Gerçeker, Binay, et al. (2018). The Child fear scale is used by the child, parent, or researcher toassess children's fear levels. The Child fear scale can be administered to measure the level of fear experienced bychildren and anxiety levels of parents for their children before, during and after procedures. This self-report scale consists of a row offive faces ranging from a'no fear neutral face'on the far left to'a faceshowing extreme fear'on the far right. The face scored '0' indicates no fear, the face scored '1' indicates a little fear, the face scored '2' indicates some fear, the face scored '3' indicates more fear and the face scored '4' indicates extreme fear.
Determining the preoperative fear scores of children | in the preoperative period.
  It assesses children's anxiety in clinical settings and uses before medical procedures. Psychometric properties of Children's anxiety meter ( in Turkish population were conducted by Gerçeker, Ayar, et al. (2018). The Children's anxiety meter (visual scale resembles a thermometer with alight bulb shape at the bottom and ten horizontal lines running from the bottom to the top. This scale is a self-report scale. A possible score that can be obtained from the Children's anxiety meter (can vary between '0' and '10'. To measure children's state anxiety levels, they are asked to mark how they feel' at the moment they are administered the Children's anxiety meter. We will measure the state anxiety levels of the children to determine their preoperative anxiety levels.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Manisa Hafsa Sultan Hospital, Manisa
  - Surgical clinic of Manisa Celal Bayar University Hospital, Manisa

REFERENCES:
- [Derived] Sekeler A, Karaarslan D, Gulmez FB. Effects of reading augmented reality storybook versus normal storybook reading on preoperative fear and anxiety levels of children in the age group of 7-12 years: A randomized controlled trial. J Pediatr Urol. 2025 Oct;21(5):1295-1305. doi: 10.1016/j.jpurol.2025.02.025. Epub 2025 Feb 25. PMID 40074655